CLINICAL TRIAL: NCT04033718
Title: Inpatient Package to Reduce HIV and AIDS-related Death in Zambia
Acronym: IPADZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University Teaching Hospital (Unknown); University of Maryland (Other)
Responsible Party: Principal Investigator, Michael Vinikoor, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 300003461
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: HIV/AIDS; Transitions of Care; Hospitalization; Tuberculosis; HIV Testing; Cryptococcosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis; Cryptococcosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient lab bundling plus navigation (Experimental): Testing for CD4 count, tuberculosis, cryptococcus, and HIV RNA with samples collected in a bundle-type approach. Additional inpatient support from a patient navigator
  Interventions: Diagnostic Test: Inpatient lab bundling; Behavioral: Inpatient navigation
- Inpatient lab bundling alone (Experimental): Testing for CD4 count, tuberculosis, cryptococcus, and HIV RNA with samples collected in a bundle-type approach.
  Interventions: Diagnostic Test: Inpatient lab bundling

INTERVENTIONS:
Diagnostic Test: Inpatient lab bundling — The investigators will provide patients a package of diagnostic tests at the time of admission to comprehensively assess for HIV coinfections and treatment failure. These labs are all recommended in advanced HIV guidelines but in this study we will provide all tests as a bundle rather than step-by-step as suggested in guidelines.
Behavioral: Inpatient navigation — Participants will be assigned a patient navigator who will support the patient and bedsider (treatment supporter/guardian) during the hospitalization. The navigator will be an HIV counselor who can provide counseling and health education, as well as support specimen transport, obtaining results, booking tests in other departments, linkages to ART clinic, and discharge planning
  Arms: Inpatient lab bundling plus navigation

SUMMARY:
Early post-discharge mortality is high among HIV-infected Zambians admitted to the hospital. Likely this is in part due to missed opportunities to identify lethal coinfections and optimize HIV care during admission (and before discharge). In this study the investigators will develop and pilot a new approach to inpatient HIV care that follows international guidelines for management of advanced HIV disease.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* HIV-positive (by self-report or DCT result in UTH file)
* Resident of Lusaka
* Admitted to the hospital

Exclusion Criteria:

* Too sick to provide informed consent (based on clinician opinion)
* Likely to be discharged in the next 48 hours (based on clinician opinion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Coinfection diagnosis | Through hospital discharge, an average of 2 weeks
  Positive test for tuberculosis or cryptococcus on admission

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Vinikoor, MD, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No